CLINICAL TRIAL: NCT01132690
Title: A Multicenter, Double-blind, Randomized Safety and Efficacy Study of Two Dose Levels of Taliglucerase Alfa in Pediatric Subjects With Gaucher Disease
Brief Title: A Safety and Efficacy Study of Two Dose Levels of Taliglucerase Alfa in Pediatric Subjects With Gaucher Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-06-005
Expanded Access: NCT00962260 (No longer available)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-09

CONDITIONS: Gaucher Disease
Keywords: gaucher disease; pediatric
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 units/kg (Experimental)
  Interventions: Drug: Taliglucerase alfa
- 60 units/kg (Experimental)
  Interventions: Drug: Taliglucerase alfa

INTERVENTIONS:
Drug: Taliglucerase alfa — Taliglucerase alfa for infusion every two weeks for 12 months
  Other Names: prGCD, plant cell expressed glucocerebrosidase

SUMMARY:
This is a multi-center, double-blind trial to assess the safety and efficacy of taliglucerase alfa in untreated subjects (2 to <18 years old) with Gaucher disease randomly assigned to treatment with one of two doses, 30 or 60 units/kg. Subjects will receive an intravenous (IV) infusion of taliglucerase alfa every two weeks. The total duration of treatment will be 12 months. At the end of the 12-month treatment period eligible subjects will be offered enrollment in an open-label extension study if taliglucerase alfa is not commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 2 to <18 years old.
* Diagnosis of Gaucher disease with leukocyte acid β-glucosidase activity ≤30% of the mean of the reference range for healthy subjects.
* Subjects who have not received enzyme replacement therapy (ERT) in the past or who have not received ERT in the past 12 months and have a negative anti-glucocerebrosidase antibody assay.
* Subjects who have not received substrate reduction therapy (SRT) in the past 12 months.
* Subjects whose clinical condition, in the opinion of the investigator, requires treatment with enzyme replacement therapy (ERT).

Exclusion Criteria:

* Currently taking another investigational drug for any condition.
* Presence of neurological signs and symptoms characteristic of Gaucher disease with complex neuronopathic features other than longstanding oculomotor gaze palsy.
* Presence of unresolved anemia due to iron, folic acid, or vitamin B12 deficiency
* Previous hypersensitivity reaction to Cerezyme® (imiglucerase) or Ceredase® (alglucerase).
* History of allergy to carrots.
* Presence of HIV, HBsAg or hepatitis C infections.
* Subject's parent(s) or legal guardian(s) are unable to understand the nature, scope and possible consequences of the study.
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the subject's compliance with the requirements of the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Shaare Zedek Medical Center, Jerusalem, Israel
- Instituto Privado de Hematologia E Investigacion Clinica (I.P.H.I.C), Barrio Sajonia Asunción, Paraguay
- Morningside Medi-Clinic, Morningside, South Africa

REFERENCES:
- [Derived] Zimran A, Gonzalez-Rodriguez DE, Abrahamov A, Elstein D, Paz A, Brill-Almon E, Chertkoff R. Safety and efficacy of two dose levels of taliglucerase alfa in pediatric patients with Gaucher disease. Blood Cells Mol Dis. 2015 Jan;54(1):9-16. doi: 10.1016/j.bcmd.2014.10.002. Epub 2014 Nov 7. PMID 25453586

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 30 Units/kg | 60 Units/kg
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30 Units/kg | 60 Units/kg | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (4.0) | 6.6 (3.1) | 8.2 (3.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Paraguay | 3 | 1 | 4
  South Africa | 1 | 2 | 3
  Israel | 2 | 2 | 4
Religion [Number; unit: participants]
  Jewish - Ashkenazi | 0 | 2 | 2
  Jewish - Non-Ashkenazi | 0 | 0 | 0
  Non Jewish | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin
Description: median and interquartile range for change from baseline in haemoglobin
Time Frame: Every 3 months for 12 months
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | 30 Units/kg | 60 Units/kg
Number analyzed (Participants) | 6 | 5
g/dL
  Month 3 | 1.2 [-0.3 to 1.6] | 0.4 [-0.1 to 1.1]
  Month 6 | 1.1 [0.3 to 2.3] | 1.5 [1.0 to 1.7]
  Month 9 | 0.9 [0.5 to 1.9] | 1.5 [1.4 to 1.6]
  Month 12 | 1.4 [0.2 to 2.5] | 1.6 [1.4 to 2.0]

2. Secondary Outcome: Chitotriosidase
Description: Percent change from baseline in chitotriosidase
Time Frame: Every 3 months for 12 months
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | 30 Units/kg | 60 Units/kg
Number analyzed (Participants) | 6 | 5
Percent Change from Baseline
  Month 3 | -32.4 (23.5) | -32.7 (15.1)
  Month 6 | -49.6 (19.8) | -50.2 (23.7)
  Month 9 | -57.2 (18.7) | -58.9 (21.8)
  Month 12 | -58.5 (17.5) | -66.1 (20.1)

3. Secondary Outcome: Spleen Volume
Description: Spleen volume measured by MRI
Time Frame: Baseline and Month 12
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 30 Units/kg | 60 Units/kg
Number analyzed (Participants) | 6 | 5
mL
  Baseline | 1218 (638.4) | 1023 (753.4)
  Month 12 | 811.6 (409.6) | 524.0 (281.1)

4. Secondary Outcome: Platelet Count
Description: Mean and standard deviation of platelet count per cubic mm
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: platelets per cubic mm
Arm/Group | 30 Units/kg | 60 Units/kg
Number analyzed (Participants) | 6 | 5
platelets per cubic mm
  Baseline | 162667 (71838) | 99600 (42899)
  Month 12 | 208167 (90747) | 172200 (89290)

5. Secondary Outcome: Chemokine (C-C Motif) Ligand 18 (CCL18)
Description: Percent change from baseline in CCL18
Time Frame: Every 3 months for 12 months
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | 30 Units/kg | 60 Units/kg
Number analyzed (Participants) | 6 | 5
Percent Change from Baseline
  Month 3 | -31.4 (15.3) | -18.3 (16.3)
  Month 6 | -45.7 (11.9) | -37.3 (28.8)
  Month 9 | -49.9 (13.0) | -46.5 (22.4)
  Month 12 | -50.6 (19.4) | -52.6 (22.5)

6. Secondary Outcome: Liver Volume
Description: Liver volume measured by MRI
Time Frame: Baseline and Month 12
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 30 Units/kg | 60 Units/kg
Number analyzed (Participants) | 6 | 5
mL
  Baseline | 1214 (424.7) | 991.7 (301.3)
  Month 12 | 1116 (366.9) | 849.1 (271.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 30 Units/kg | 60 Units/kg
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 2/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 Units/kg (N=6) | 60 Units/kg (N=5)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 Units/kg (N=6) | 60 Units/kg (N=5)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No